CLINICAL TRIAL: NCT04500730
Title: Effectiveness of Herbal Medicine (Shaoyao Gancao Decoction Jiawei) in Sleep-related Leg Cramps - A Pilot Study
Brief Title: Evaluate the Efficacy of Herbal Medicine (Shaoyao Gancao Decoction Jiawei) in Sleep-related Leg Cramps
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Chinese University of Hong Kong (Other)
Responsible Party: Principal Investigator, Prof. Lin Zhixiu, Associate professor, Chinese University of Hong Kong
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SRLC study
Record Dates: First submitted 2020-08-03; First posted 2020-08-05 (Actual); Last update posted 2020-08-28 (Actual); Status verified 2020-08

CONDITIONS: Sleep-related Leg Cramps

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Shaoyao Gancao Decoction Jiawei (Experimental): Shaoyao Gancao Decoction Jiawei by adding Pueraria montana, Salvia Miltiorrhiza, into Shaoyao Gancao.
  The medication will be taken twice daily for 28 consecutive days. Each prescription will consist of 4 herbal granules.
  Interventions: Drug: Shaoyao Gancao Decoction Jiawei

INTERVENTIONS:
Drug: Shaoyao Gancao Decoction Jiawei — Study herb will be prescribed for 28 consecutive days. Study follow up will be offered every 7 days till 56th day after enrolment.
  Daily leg cramps log will be filled in by each individual everyday from day 0 to day 56.
  Other Names: Nong's Concentrated Chinese Medicine Granules

SUMMARY:
Sleep-related leg cramps (SRLCs) are a sleep-related movement disorder whereby painful contractions of the calf or foot muscles arise at sleep onset and during sleep and awaken the patient, interrupting sleep. Application of oral administration with Chinese herbal medicine can enhance the effectiveness and efficacy in treatment of SRLCs.This study will using Shaoyao Gancao Prescription Jiawei by adding Pueraria montana, Salvia Miltiorrhiza, into Shaoyao Gancao. The study aims to evaluate the effectiveness of a Shaoyao Gancao Prescription Jiawei in relieving leg cramps.

DETAILED DESCRIPTION:
The study will be conducted in Yan Oi Tong Mrs Shirley W K Siu Medical Centre. All participants diagnosed with sleep-related leg cramp will be screened for eligibility criteria from the general public or referred patients via daily outpatient services. This will be a prospective trial in patients with sleep-related leg cramps (SRLCs). 30 subjects will be recruited from Yan Oi Tong Mrs Shirley W K Siu Medical Centre. The medication will be taken twice daily for 28 consecutive days. Each prescription will consist of 4 herbal granules. Study follow up will be offered every 7 days till 56th day after enrolment. Daily leg cramps log will be filled in by each individual everyday from day 0 to day 56.

ELIGIBILITY:
Inclusion Criteria:

1. Aged 60-80
2. Complain of muscular spasm and contracture of a limb with difficulty in relaxation and movement during night time, caused by wind-cold dampness chiefly involving the sinews
3. SRLCs occur at least once in the past 7 days or twice in the past 14 days
4. Visual Analogue Scale (VAS) for leg cramp ≥ 5 (0-10) at the last attack
5. Both gender but menopause or sterilization for female subjects
6. Able to fill up the VAS for leg cramp
7. Written informed consent obtained

Exclusion Criteria:

1. Known mental disorder 2. Known serious organic disease including severe coronary function impairment, post-stroke depression and dementia, and auto-immune diseases 3. Known history of renal or liver function impairment; 4. Patients whose blood tests show exclusion criteria 5. Currently taking anticoagulant or antiplatelet 6. Any contraindications for taking herb confirmed by investigator

-

Ages: 60 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2019-08-01 (Actual); Primary Completion 2019-12-31 (Actual); Study Completion 2019-12-31 (Actual)

PRIMARY OUTCOMES:
Visual Analogue Score (VAS) Assessment | 4 Weeks
  The pain VAS is a unidimensional measure of pain intensity, it ranges from 0 to 10cm,high score means more painful.

SECONDARY OUTCOMES:
Short Form 36 Health Survey Questionnaire | 8 weeks
  to assess the health-related quality of life of subjects, it ranges from 0-100 scores, the higher the score, the more disability
Visual Analogue Score (VAS) Assessment | 8 weeks
  The pain VAS is a unidimensional measure of pain intensity, it ranges from 0 to 10cm,high score means more painful.

CONTACTS AND LOCATIONS:
Locations (1):
- The Chinese University of Hong Kong, Hong Kong, Hong Kong